CLINICAL TRIAL: NCT00234130
Title: A Comparison of the Effects of Conventional and Nocturnal Hemodialysis on the Inflammatory Response of Chronic Renal Failure
Brief Title: The Effect of Nighttime Dialysis on the Inflammation of Kidney Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient population was not enough to complete enrollment
Sponsor: Rockefeller University (Other)
Collaborators: The Rogosin Institute (Other)
Responsible Party: Lisa Hudgins, MD, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUH IRB # LHU 0486
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: End-Stage Renal Disease
Keywords: Dialysis; Cytokines; Triglycerides; Insulin
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: nocturnal vs conventional dialysis

SUMMARY:
This study will determine whether a new form of home hemodialysis carried out at night during sleep reduces blood levels of hormone-like substances called cytokines that may cause fatigue and increase blood fats and sugar. Participants will stay twice in the Rockefeller Hospital and receive a standard diet and blood testing. Training for nocturnal hemodialysis will be provided at the nearby Manhattan Dialysis Center of The Rogosin Institute, affiliated with The Rockefeller University.

DETAILED DESCRIPTION:
Patients treated with conventional hemodialysis for at least 3 months and interested in learning home nocturnal hemodialysis will be screened in the Rockefeller Outpatient Research Center. If eligible, during the first 8 day hospital stay, participants will receive a standard diet and dialysis treatment nearby at the Rogosin Institute Dialysis Center. During the last 2 days, their blood will be frequently sampled for cytokines, fats and sugar. Dialysate will also be sampled. They will have the same diet and tests repeated during a second admission after either 4 months of conventional dialysis or 1 month training for nocturnal dialysis followed by 3 months of home nocturnal dialysis (randomized 1:1). After the second admission, patients treated with conventional dialysis will be discharged from the study and trained in nocturnal hemodialysis. Off-site computer monitoring will be utilized when patients dialyze themselves at home or during the admission in The Rockefeller University Hospital.

ELIGIBILITY:
Inclusion Criteria:

Men and women at least age 18 who receive hemodialysis three times a week for at least 3 months and meet the criteria for home instruction in nocturnal dialysis -

Exclusion Criteria:

No diabetes, any unstable clinical condition, chronic infection (including hepatitis, HIV), endocrine disorders or serious digestive problems, lipid-lowering medication , LDL cholesterol <190 mg/dL and triglycerides less than 600 mg/dL, body mass index <35, blood pressure <160/100, hemoglobin >10.0, no cholesterol-lowering medicine, able to change from Renagel (has lipid effects) to Phoslo for the duration of the study, cigarette smoking no more than half a pack per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Feasibility study

SECONDARY OUTCOMES:
Feasibility study

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C. Hudgins, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.rucares.org/clinicalstudies/list.php